CLINICAL TRIAL: NCT04530240
Title: Impact of National MELD ≥ 30 Priority Allocation System on Dropout and Post-Transplant Survival Rates in Italy: A Retrospective Competing-Risk Analysis
Brief Title: Equity and Efficacy of Allocation Priority for Liver Transplantation Patients With MELD≥30 in Italy
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Collaborators: University of Roma La Sapienza (Other); University of Pisa (Other); A.O.U. Città della Salute e della Scienza (Other); Niguarda Hospital (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Matteo Ravaioli, Professor, Professor, University of Bologna
Other Study IDs: Reg.Pg284644
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Liver Transplant Disorder; HCC
Keywords: Allocation System; Liver Transplantation
MeSH Terms: interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ERA-1 Group: Before the introduction of the MELD≥30 allocation scheme August 2010 - July 2014
  Interventions: Procedure: Liver Transplantation
- ERA-2 Group: After the introduction of the MELD≥30 allocation scheme August 2014 - July 2018
  Interventions: Procedure: Liver Transplantation

INTERVENTIONS:
Procedure: Liver Transplantation — Use prospectively collected databases from each participate centre, register MELD score recorded at the time of drop-out, liver transplantation and end of the follow-up.

SUMMARY:
In Italy, since August 2014, liver transplantation (LT) candidates with MELD≥30 receive a priority allocation consenting them to access in an organ sharing macroarea. The primary intent of this policy is to minimize the higher risk of waiting list dropout observed in these patients. Another objective of this allocation strategy is to reduce the waiting time, thus performing the LT in better clinical conditions. This multicentre retrospective national study aims to evaluate several parameters of efficacy and equity, such as waiting time in the list, dropout rate, and graft survival, in two eras of enlisted patients, before and after the introduction of the macroarea sharing policy in Italy. With the intent to minimize the presence of possible selection biases, the two groups were matched trough Propensity Score Matching (PSM).

DETAILED DESCRIPTION:
A retrospective multi-centre study involving six Italian transplant centres was performed using prospectively collected databases from each participating centre, registering MELD score recorded at the time of drop-out, liver transplantation and end of the follow-up.

Study population was divided in two groups according to the time of waiting list before or after the introduction of MELD ≥ 30 allocation scheme: ERA-1 Group (August 2010 - July 2014), and ERA-2 Group (August 2014 - July 2018).

Primary endpoint was waiting list time across different eras in patients above and below MELD ≥ 30 cutoff. Secondary endpoints were dropout rate as well as patient and graft survival.

ELIGIBILITY:
Inclusion Criteria:

- LT patients registered from August 2010 to July 2018

Exclusion Criteria:

* LT patients registered before August 2010 and after July 2018
* Data not available for analysis

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 4,238 LT patients registered from August 2010 to July 2018 have been initially enrolled for the analysis (Bologna=961, Pisa=980, Turin=897, Milan Niguarda=859, Rome Sapienza=268, Rome Cattolica=273), and categorized in an ERA-1 Group (n=2,225; before macroarea priority allocation), and an ERA-2 Group (n=2,013; after macroarea priority allocation).
Sampling Method: Non-Probability Sample
Enrollment: 4238 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Patient Survival | 5 year
  Survival since waiting list and after liver transplantation

SECONDARY OUTCOMES:
Graft Survival | 5 year
  Survival of the graft since liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Ravaioli, Professor, Principal Investigator — Sant'Orsola-Malpighi Hospital, University of Bologna

REFERENCES:
- [Background] Ravaioli M, Grazi GL, Ballardini G, Cavrini G, Ercolani G, Cescon M, Zanello M, Cucchetti A, Tuci F, Del Gaudio M, Varotti G, Vetrone G, Trevisani F, Bolondi L, Pinna AD. Liver transplantation with the Meld system: a prospective study from a single European center. Am J Transplant. 2006 Jul;6(7):1572-7. doi: 10.1111/j.1600-6143.2006.01354.x. PMID 16827857
- [Background] Kamath PS, Wiesner RH, Malinchoc M, Kremers W, Therneau TM, Kosberg CL, D'Amico G, Dickson ER, Kim WR. A model to predict survival in patients with end-stage liver disease. Hepatology. 2001 Feb;33(2):464-70. doi: 10.1053/jhep.2001.22172. PMID 11172350
- [Background] Nekrasov V, Matsuoka L, Rauf M, Kaur N, Cao S, Groshen S, Alexopoulos SP. National Outcomes of Liver Transplantation for Model for End-Stage Liver Disease Score >/=40: The Impact of Share 35. Am J Transplant. 2016 Oct;16(10):2912-2924. doi: 10.1111/ajt.13823. Epub 2016 May 13. PMID 27063579
- [Background] Goldberg DS, Levine M, Karp S, Gilroy R, Abt PL. Share 35 changes in center-level liver acceptance practices. Liver Transpl. 2017 May;23(5):604-613. doi: 10.1002/lt.24749. PMID 28240804
- [Background] Weismuller TJ, Fikatas P, Schmidt J, Barreiros AP, Otto G, Beckebaum S, Paul A, Scherer MN, Schmidt HH, Schlitt HJ, Neuhaus P, Klempnauer J, Pratschke J, Manns MP, Strassburg CP. Multicentric evaluation of model for end-stage liver disease-based allocation and survival after liver transplantation in Germany--limitations of the 'sickest first'-concept. Transpl Int. 2011 Jan;24(1):91-9. doi: 10.1111/j.1432-2277.2010.01161.x. Epub 2010 Sep 3. PMID 20819196
- [Background] Habib S, Berk B, Chang CC, Demetris AJ, Fontes P, Dvorchik I, Eghtesad B, Marcos A, Shakil AO. MELD and prediction of post-liver transplantation survival. Liver Transpl. 2006 Mar;12(3):440-7. doi: 10.1002/lt.20721. PMID 16498643
- [Background] Nicolas CT, Nyberg SL, Heimbach JK, Watt K, Chen HS, Hathcock MA, Kremers WK. Liver transplantation after share 35: Impact on pretransplant and posttransplant costs and mortality. Liver Transpl. 2017 Jan;23(1):11-18. doi: 10.1002/lt.24641. Epub 2016 Dec 5. PMID 27658200
- [Background] Ravaioli M, Grande G, Di Gioia P, Cucchetti A, Cescon M, Ercolani G, Del Gaudio M, Morelli C, Pinna AD. Risk Avoidance and Liver Transplantation: A Single-center Experience in a National Network. Ann Surg. 2016 Nov;264(5):778-786. doi: 10.1097/SLA.0000000000001887. PMID 27429038
- [Background] Nagai S, Chau LC, Schilke RE, Safwan M, Rizzari M, Collins K, Yoshida A, Abouljoud MS, Moonka D. Effects of Allocating Livers for Transplantation Based on Model for End-Stage Liver Disease-Sodium Scores on Patient Outcomes. Gastroenterology. 2018 Nov;155(5):1451-1462.e3. doi: 10.1053/j.gastro.2018.07.025. Epub 2018 Jul 26. PMID 30056096
- [Background] Kwong AJ, Goel A, Mannalithara A, Kim WR. Improved posttransplant mortality after share 35 for liver transplantation. Hepatology. 2018 Jan;67(1):273-281. doi: 10.1002/hep.29301. Epub 2017 Nov 13. PMID 28586179
- [Background] Beal EW, Black SM, Mumtaz K, Hayes D Jr, El-Hinnawi A, Washburn K, Tumin D. High Center Volume Does Not Mitigate Risk Associated with Using High Donor Risk Organs in Liver Transplantation. Dig Dis Sci. 2017 Sep;62(9):2578-2585. doi: 10.1007/s10620-017-4639-2. Epub 2017 Jun 1. PMID 28573507
- [Background] Kang S, Little RJ, Kaciroti N. Missing not at random models for masked clinical trials with dropouts. Clin Trials. 2015 Apr;12(2):139-48. doi: 10.1177/1740774514566662. Epub 2015 Jan 27. PMID 25627429
- [Background] Caliendo M, Kopeinig S. Some practical guidance for the implementation of propensity score matching. J Econ Surv. 2008; 22:31-72
- [Background] Austin PC, Lee DS, Fine JP. Introduction to the Analysis of Survival Data in the Presence of Competing Risks. Circulation. 2016 Feb 9;133(6):601-9. doi: 10.1161/CIRCULATIONAHA.115.017719. PMID 26858290
- [Background] Nekrasov V, Matsuoka L, Kaur N, Pita A, Whang G, Cao S, Groshen S, Alexopoulos S. Improvement in the Outcomes of MELD >/= 40 Liver Transplantation: An Analysis of 207 Consecutive Transplants in a Highly Competitive DSA. Transplantation. 2017 Oct;101(10):2360-2367. doi: 10.1097/TP.0000000000001738. PMID 28319564
- [Background] Luo X, Leanza J, Massie AB, Garonzik-Wang JM, Haugen CE, Gentry SE, Ottmann SE, Segev DL. MELD as a metric for survival benefit of liver transplantation. Am J Transplant. 2018 May;18(5):1231-1237. doi: 10.1111/ajt.14660. Epub 2018 Feb 19. PMID 29316310
- [Background] Ravaioli M, Grazi GL, Ercolani G, Cescon M, Del Gaudio M, Zanello M, Ballardini G, Varotti G, Vetrone G, Tuci F, Lauro A, Ramacciato G, Pinna AD. Liver allocation for hepatocellular carcinoma: a European Center policy in the pre-MELD era. Transplantation. 2006 Feb 27;81(4):525-30. doi: 10.1097/01.tp.0000198741.39637.44. PMID 16495798
- [Background] Ghinolfi D, Lai Q, Pezzati D, De Simone P, Rreka E, Filipponi F. Use of Elderly Donors in Liver Transplantation: A Paired-match Analysis at a Single Center. Ann Surg. 2018 Aug;268(2):325-331. doi: 10.1097/SLA.0000000000002305. PMID 28549011
- [Background] Cillo U, Burra P, Mazzaferro V, Belli L, Pinna AD, Spada M, Nanni Costa A, Toniutto P; I-BELT (Italian Board of Experts in the Field of Liver Transplantation). A Multistep, Consensus-Based Approach to Organ Allocation in Liver Transplantation: Toward a "Blended Principle Model". Am J Transplant. 2015 Oct;15(10):2552-61. doi: 10.1111/ajt.13408. Epub 2015 Aug 14. PMID 26274338
- [Background] Sundaram V, Kogachi S, Wong RJ, Karvellas CJ, Fortune BE, Mahmud N, Levitsky J, Rahimi RS, Jalan R. Effect of the clinical course of acute-on-chronic liver failure prior to liver transplantation on post-transplant survival. J Hepatol. 2020 Mar;72(3):481-488. doi: 10.1016/j.jhep.2019.10.013. Epub 2019 Oct 25. PMID 31669304
- [Background] Jasseron C, Francoz C, Antoine C, Legeai C, Durand F, Dharancy S; collaborators. Impact of the new MELD-based allocation system on waiting list and post-transplant survival - a cohort analysis using the French national CRISTAL database. Transpl Int. 2019 May 10. doi: 10.1111/tri.13448. Online ahead of print. PMID 31074921
- [Background] Tschuor C, Ferrarese A, Kuemmerli C, Dutkowski P, Burra P, Clavien PA; Liver Allocation Study Group. Allocation of liver grafts worldwide - Is there a best system? J Hepatol. 2019 Oct;71(4):707-718. doi: 10.1016/j.jhep.2019.05.025. Epub 2019 Jun 12. PMID 31199941
- [Background] Ishaque T, Massie AB, Bowring MG, Haugen CE, Ruck JM, Halpern SE, Waldram MM, Henderson ML, Garonzik Wang JM, Cameron AM, Philosophe B, Ottmann S, Rositch AF, Segev DL. Liver transplantation and waitlist mortality for HCC and non-HCC candidates following the 2015 HCC exception policy change. Am J Transplant. 2019 Feb;19(2):564-572. doi: 10.1111/ajt.15144. Epub 2018 Nov 9. PMID 30312530
- [Background] Yoo S, Jang EJ, Yi NJ, Kim GH, Kim DH, Lee H, Jung CW, Ryu HG. Effect of Institutional Case Volume on In-hospital Mortality After Living Donor Liver Transplantation: Analysis of 7073 Cases Between 2007 and 2016 in Korea. Transplantation. 2019 May;103(5):952-958. doi: 10.1097/TP.0000000000002394. PMID 30086090
- [Derived] Ravaioli M, Lai Q, Sessa M, Ghinolfi D, Fallani G, Patrono D, Di Sandro S, Avolio A, Odaldi F, Bronzoni J, Tandoi F, De Carlis R, Pascale MM, Mennini G, Germinario G, Rossi M, Agnes S, De Carlis L, Cescon M, Romagnoli R, De Simone P. Impact of MELD 30-allocation policy on liver transplant outcomes in Italy. J Hepatol. 2022 Mar;76(3):619-627. doi: 10.1016/j.jhep.2021.10.024. Epub 2021 Nov 10. PMID 34774638